CLINICAL TRIAL: NCT02204501
Title: A Phase 1, Randomized, Open-Label Study to Evaluate the Effect of Vapendavir (BTA798) on the Pharmacokinetics of Orally Administered Midazolam, a CYP3A4 Substrate, in Healthy Male and Female Volunteers
Brief Title: A Drug-Drug Interaction Study to Evaluate the Effect of Vapendavir on the Pharmacokinetics of Midazolam in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biota Scientific Management Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BTA798-102
Record Dates: First submitted 2014-05-27; First posted 2014-07-30 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Drug-Drug Interaction Healthy Volunteers
Keywords: Aviragen Therapeutics, Inc.; Aviragen Therapeutics; Aviragen
MeSH Terms: interventions — Midazolam; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vapendavir 528 mg QD (Experimental): Twelve subjects (6 male and 6 female) will receive 528 mg vapendavir (achieved with four 132 mg vapendavir capsules) QD in the morning for seven days
  Interventions: Drug: Midazolam 5mg Syrup; Drug: Vapendavir 528 mg QD
- Vapendavir 264 mg BID (Experimental): Twelve subjects (6 male and 6 female) will receive 264 mg vapendavir (achieved with two 132 mg vapendavir capsules) BID daily as divided dose given in the morning and evening 12 hours apart for seven days.
  Interventions: Drug: Midazolam 5mg Syrup; Drug: Vapendavir 264 mg BID

INTERVENTIONS:
Drug: Midazolam 5mg Syrup — All twenty four subjects will receive 5 mg midazolam syrup at four different time points during the study for a total of four non-subsequent dosing days.
  * On Study Days 0 and 12, subjects will receive only 5 mg midazolam syrup dosed in the morning.
  * On Study Days 6 and 9, subjects will have 5 mg midazolam syrup co-administered with their assigned dose of vapendavir in the morning. Co-administration of midazolam will not occur at the time of the evening dose for Group B.
Drug: Vapendavir 264 mg BID — Twelve subjects (6 male and 6 female) will receive 264 mg vapendavir (achieved with two 132 mg vapendavir capsules) BID daily as divided dose given in the morning and evening 12 hours apart for seven days.
  Arms: Vapendavir 264 mg BID
Drug: Vapendavir 528 mg QD — Twelve subjects (6 male and 6 female) will receive 528 mg vapendavir (achieved with four 132 mg vapendavir capsules) QD in the morning for seven days
  Arms: Vapendavir 528 mg QD

SUMMARY:
The primary aim of this Phase 1 study is to evaluate the effect of vapendavir daily doses of 528 mg daily (QD) and 264 mg twice daily (BID) on the pharmacokinetic (PK) profile of midazolam, a cytochrome (CYP) 3A4 substrate. Additionally, the effect of midazolam on the PK profile of vapendavir, a PK profile comparison of vapendavir in males and females, as well as the safety of vapendavir will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female between 18 and 55 years of age (inclusive) with BMI between 18 and 30 kg/m2 (inclusive), and weight ≥50 kg at the time of screening;
* Capable of giving written informed consent;
* Subject is able to understand and comply with the protocol requirements, instructions and restrictions;
* Healthy on the basis of physical examination, medical history, medication usage, vital signs (VS), electrocardiograms (ECGs), and clinical laboratory tests;
* Female subjects who are not post-menopausal for at least 2 years or surgically sterile with complete hysterectomy or bilateral oophorectomy and male subjects who are not surgically sterile via vasectomy, must agree to use a double barrier method of birth control, such as a condom plus spermicidal agent (foam/gel/film/cream/suppository); and
* Female subjects must not be breastfeeding or pregnant.

Exclusion Criteria:

* Positive results for Hepatitis B, Hepatitis C, or HIV;
* Frequent use (defined as > 5 times/day) of tobacco products, including cigarettes, cigars, chewing tobacco;
* A medical history of significant hematological, gastrointestinal, respiratory, renal, hepatic, cerebrovascular, immunologic, psychiatric or cardiovascular disease or event;
* Current or recent respiratory infection (defined as within 14 days of first study visit participation)
* Presence or history of significant allergy;
* Clinically significant abnormalities noted on ECG;
* Screening vital signs representing sustained elevated systolic blood pressure <90 mmHg or >140 mmHg, and/or diastolic blood pressure <55 mmHg or >90 mmHg.
* Presence of significant gastrointestinal abnormalities such as diarrhea or constipation;
* Safety laboratory abnormalities noted at screening which are clinically significant
* Current or defined history of abuse of alcohol or illicit drugs;
* A positive pregnancy test at screening;
* Poor vein access or fear of venipuncture or sight of blood; and
* Regular consumption of alcohol defined as either > 2 units (glass or shot) of alcoholic beverages per day or > 14 units per week.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The Effect of Vapendavir on the PK Profile of Midazolam | End of Study (up to 46 weeks in duration)
  To evaluate the effect of vapendavir daily dose of 264 mg BID on the PK profile of midazolam, a CYP3A4 substrate. The primary outcome will be evaluated through a series of analyses of PK parameters including:
  * for midazolam including maximum observed plasma concentration (Cmax)
  * time at which Cmax was observed (Tmax)
  * plasma concentration at the end of the dosing interval (Ctau)
  * area under the plasma concentration-time curve from time 0 to the last measurable plasma concentration (AUC0-last)
  * area under the plasma concentration-time curve from time 0 to the end of the dosing interval (AUC0-tau)
  * area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-inf)
  * elimination half-life (t1/2)
  * apparent oral clearance (CL/F)
  * apparent oral volume of distribution (Vz/F).
The Effect of Vapendavir on the PK Profile of Midazolam | End of Study (up to 46 weeks in duration)
  To evaluate the effect of vapendavir daily dose of 528 mg QD on the PK profile of midazolam, a CYP3A4 substrate. The primary outcome will be evaluated through a series of analyses of PK parameters including:
  * for midazolam including maximum observed plasma concentration (Cmax)
  * time at which Cmax was observed (Tmax)
  * plasma concentration at the end of the dosing interval (Ctau)
  * area under the plasma concentration-time curve from time 0 to the last measurable plasma concentration (AUC0-last)
  * area under the plasma concentration-time curve from time 0 to the end of the dosing interval (AUC0-tau)
  * area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-inf)
  * elimination half-life (t1/2)
  * apparent oral clearance (CL/F)
  * apparent oral volume of distribution (Vz/F).

SECONDARY OUTCOMES:
Assess Whether PK Profile of Vapendavir is Affected by Presence of Midazolam | End of Study (up to 46 weeks in duration)
  To evaluate whether the PK profile of vapendavir, is affected by the presence of midazolam, a strong CYP3A4 substrate. This outcome will be evaluated through a series of analyses of PK parameters for vapendavir including:
  * maximum observed plasma concentration (Cmax)
  * time at which Cmax was observed (Tmax)
  * plasma concentration at the end of the dosing interval (Ctau)
  * area under the plasma concentration-time curve from time 0 to the last measurable plasma concentration (AUC0-last)
  * area under the plasma concentration-time curve from time 0 to the end of the dosing interval (AUC0-tau)
  * area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-inf)
  * elimination half-life (t1/2)
  * apparent oral clearance (CL/F)
  * apparent oral volume of distribution (Vz/F).
Assess the Safety of Vapendavir | End of Study (up to 46 weeks in duration
  To evaluate the safety of vapendavir. This will be accomplished by assessing adverse events, clinical laboratory tests (including blood chemistry, hematology with differential and urinalysis), physical exams, ECG assessments, vital sign assessments and concomitant medications.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Matson, MD, Principal Investigator — Prism Clinical Research
Locations (1):
- Prism Clinical Research, Saint Paul, Minnesota, United States